CLINICAL TRIAL: NCT05864287
Title: Pac-12 Test of the Effectiveness of Bodies in Motion in Reducing Disordered Eating and Body Image Concerns, and Improving Psychological Well-Being, Among Male and Female Student-Athletes
Brief Title: Pac-12 Test of the Effectiveness of Bodies in Motion in Reducing Disordered Eating and Body Image Concerns
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: University of North Texas Health Science Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000865
Record Dates: First submitted 2022-09-30; First posted 2023-05-18 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2024-08

CONDITIONS: Effectiveness of BIM in Reducing Disordered Eating Among Student Athletes; Effectiveness of BIM in Reducing Body Image Concerns Among Student Athletes; Effectiveness of BIM Improving Psychological Well-Being Among Student Athletes

STUDY DESIGN:
Intervention Model Description: No treatment control
Masking Description: This is an open trial of Bodies In Motion (BIM) Intervention. The study will primarily examine results pre-post treatment within these athletes. However, athletes who do not sign up to participate in the BIM may be used as "no treatment controls", utilizing data collected during their bi-annual mental health screens and propensity matching. However, this does not typically qualify as an "Arm".
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BIM intervention participants (Other): Specifically, at each of the seven intervention sites, a minimum of 30 male and 30 female-identifying student athletes will participate in the BIM program across the 2022-2023 academic year. Thus, our intervention sample will be a minimum of 210 male and 210 female identifying intervention group athletes. The BIM program is a manualized intervention that consists of a 35-min introductory session, followed by four, 75-min sessions. Athletes participating in BIM who give consent (via electronic consent documentation) to share their de-identified data for research purposes will complete additional surveys beyond the standard MH-CDE set of baseline measures at one time-point and treatment-related measures at five time-points:
  * Pre-intervention/Baseline
  * Post-intervention (1-2 weeks after)
  * 4-months post-intervention
  * 12-months post-intervention
  Interventions: Behavioral: Bodies in motion intervention program

INTERVENTIONS:
Behavioral: Bodies in motion intervention program — Intervention groups will be offered separately to male- and female-identifying athletes; each group will consist of six to eight athletes and multiple groups may be run each academic term. Facilitators will use the gender-specific programs in their delivery. Intervention athletes will receive a participant workbook as well as be invited to join a BIM-specific, private social media platform that will allow them to share, connect, and support each other through out their involvement in the program. As part of our mixed-methods design, we will also conduct qualitative interviews to explore the student athletes' experiences of the BIM program. Following intervention, we will invite 12-16 male and 12-16 female identifying athletes who completed the BIM program to participate in the structured interviews. Interviews will be semi-structured and are expected to last 60-90 minutes

SUMMARY:
In the proposed study, the investigators will examine the effectiveness of Bodie in Motion (BIM) program in improving the body image, eating concerns, and overall psychological well-being, in a racially/ethnically diverse group of female and male-identifying athletes with body image concerns. Based on previous research, participating athletes should have direct and immediate Well-Being (i.e., mental health) benefits from their involvement in BIM.

DETAILED DESCRIPTION:
The Primary Aim of this project is to modify (based on diverse college student athlete acceptability and effectiveness feedback) and then further test the effectiveness of the evidence-based Bodies in Motion (BIM) program in reducing the body image concerns, decreasing the disordered eating symptoms, and improving the psychological well-being (e.g., depression, anxiety) in a racially/ethnically diverse group of female and male-identifying student-athletes in the Pac-12 conference.

The primary hypothesis is that, compared to treatment as usual (TAU) control athletes who have been matched on race, ethnicity, sport, and gender (male vs. female-identifying), athletes completing the BIM treatment will have greater improvements on body image and eating concerns, and lower levels of depression and anxiety. These differences will occur immediately following completion of BIM and will be maintained at 6- and 12-months. In keeping with our mixed-methods approach, through qualitative interviews conducted with the athletes who have participated in the BIM program, the investigators will explore their perceptions of the program's efficacy, relative to how the awareness, perspectives, and skills developed from the program have, or have not, informed their relationship with themselves, their bodies, food, physical activity, and general psychological well-being. The investigators expect that, based on past research (Voelker, Petrie et al., 2021) that athletes will report increased awareness of self and body, positive shifts in how they view themselves and their bodies, and the adoption of psychological tools (e.g., mindful self-compassion) to cope more effectively with appearance stressors.

The secondary Aim is to determine if the BIM program's effectiveness differs based on athletes' race/ ethnicity within each gender (e.g., for female-identifying athletes). That is, does athlete race/ethnicity moderate their BIM outcomes.

Exploratory aims include examining if sport played and facilitators' professional training (e.g., sport nutritionist, sport psychologist) further moderate outcomes.

Student athletes will be recruited through self-selection into the Bodies in Motion (BIM) program from one of the seven participating schools who will be offering this treatment. Athletes who A) self-identify as experiencing body image concerns, or B) are referred by someone (e.g., nutritionist, athletic trainer) based on some expressed body dissatisfaction. Each university intervention site will offer BIM to its athletes as a clinical service. And upon enrolling in BIM, athletes will be presented with an overview of the ongoing research study and the opportunity to provide consent for their intervention data to be shared for research purposes. Consent to sharing data for research purposes will not be required for participating in BIM. Athletes participating in BIM who give consent to share their data for research purposes (via electronic consent documentation) will complete additional surveys related to treatment outcomes.

Once the investigators have the BIM intervention participants identified and consented into the study, the investigators will then go into the MH-CDE screener data to find "matched" participants at other schools.

Matched-control participants will already be completing the Mental Health Common Data Elements (MH-CDEs) as part of their biannual mental health screeners in their respective athletics department. As part of their clinical care within the various athletic departments, student-athletes are asked to complete a variety of assessments (e.g., physical, MH-CDEs, etc.). The MH-CDEs are currently delivered via REDCap through a link provided in email. For the matched-control participants, the investigators will have a consent at the end of the MH-CDEs explaining the study and asking if the investigators can utilize their data for research purposes. The investigators will make it clear that participating in our study (i.e., allowing us to use their data) in no way affects their ability to participate in sports.

ELIGIBILITY:
Inclusion Criteria:

* Current student-athlete
* At least 18 years of age at a Pac-12 University
* Fluently read, write, and speak English.

Exclusion Criteria:

• Unwilling to provide informed consent.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-08-08 (Actual); Study Completion 2024-08-08 (Actual)

PRIMARY OUTCOMES:
Change between baseline and post intervention Weight Pressures in Sport (WPS) Scale | pre-intervention, 1-2 weeks, 4 months and 12 months post intervention
  Self-reported weight loss pressures from the external environment.
Change between baseline and post intervention Sociocultural Attitudes Toward Appearance Questionnaire-4 (SATAQ-4 | pre-intervention, 1-2 weeks, 4 months and 12 months post intervention
  Self-reported thinness and muscularity internalization.
Change between baseline and post intervention Sociocultural Attitudes Toward Appearance Questionnaire | pre-intervention, 1-2 weeks, 4 months and 12 months post intervention
  Self-reported weight loss, thinness and muscularity perceived from outside pressures.
Change between baseline and post intervention Body Parts Satisfaction Scale-Revised (BPSS-R) | pre-intervention, 1-2 weeks, 4 months and 12 months post intervention
  Self-reported body part satisfaction
Change between baseline and post intervention Self-Compassion Scale - Short Form (SCS-SF) | pre-intervention, 1-2 weeks, 4 months and 12 months post intervention
  Self-reported frequency of self-compassionate attitudes and behaviors.

SECONDARY OUTCOMES:
Patient Health Questionnaire-2 Item (PHQ-2 | Baseline
  Self-reported frequency of depressed mood and anhedonia.
Generalized Anxiety Disorder-2 Item (GAD-2) | Baseline
  Self-reported severity of frequency of nervous/anxious/on edge/worry behaviors.
Eating Disorder Examination Questionnaire-Short Form (EDE-QS) | Baseline
  Self-reported eating disorder symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Taylor, Ph.D, Principal Investigator — University of Arizona
Locations (1):
- The university of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No